CLINICAL TRIAL: NCT06108011
Title: Effect of Lollipop on Postoperative Gastrointestinal Recovery in Children: A Randomised Controlled Trial
Brief Title: Effect of Lollipop on Postoperative Gastrointestinal Recovery in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LollipopTrial
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Ileus Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lollipop (Experimental): Given lollipop 6 hours after operation, sucking of lollipop at least 20mins every 4 hours after operation until feeding is resumed.
  Interventions: Other: Lollipop
- No Lollipop (No Intervention): No placebo would be given

INTERVENTIONS:
Other: Lollipop — sucking of lollipop after operation
  Arms: Lollipop

SUMMARY:
Postoperative ileus is common in children. There are various method to prevent postoperative ileus. In this study, the investigators will explore the role of sucking lollipop after operation on the recovery of gastrointestinal function in children.

DETAILED DESCRIPTION:
Postoperative ileus is a common occurrence among children undergoing major operations, including gastrointestinal and spinal surgeries. It can result in physical discomfort, extended hospital stays, delayed resumption of activity and poor satisfaction with surgical care. The pathophysiology and course of postoperative ileus occurs in three phases: increased sympathetic activity, release of inflammatory mediators and vagal activation as ileus resolves. Multiple risk factors of postoperative ileus have been identified in various studies, including general risk factors such as significant blood loss, male gender and medical comorbidities like chronic obstructive pulmonary disease (COPD), as well as risk factors specific to the surgery, such as the laparotomy approach, emergency surgery and stoma formation.

Chewing gum, as a form of sham feeding, has been employed in adults and children as a modality to decrease risk of postoperative ileus. There has been concrete evidence that it could result in expedited recovery of gastrointestinal function after surgery in adult populations. However, it may not be a feasible option for infants and young children. Lollipop, on the other hand, is easier to apply in children which only require the action of sucking. It can stimulate the cephalic phase of digestion via vagal cholinergic stimulation and release of gastrointestinal hormone (gastrin and motilin) through its taste and absorption of sugar. The current evidence of lollipop in the recovery of postoperative gastrointestinal function in children is limited with only two randomised controlled trial published so far with satisfactory outcomes, yet both were not indexed and were not carried out in accordance with Consolidated Standards of Reporting Trials (CONSORT). Based on these reasons, the investigators plan to carry out a prospective, multiple-centred, non-blinded, randomized controlled trial using a parallel arm design on the effect of lollipop on recovery of gastrointestinal function after operation in children. Children recruited will be randomly assigned into either lollipop group or non-treatment group; lollipop will be given to children in treatment group after operation. Their outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving major abdominal surgery (e.g.appendicectomy, choledochal cyst surgery, bowel resection etc)

Exclusion Criteria:

* Patients with neurological conditions that preclude sucking/swallowing.
* Patients under sedation and/or mechanical ventilation and/or ionotropic support in the post operative period.
* Patients with known food allergy or allergy to food coloring agents

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time for participants to return of flatus | 1 week
  the time needed for flatus to happen after operation, in term as hours
Time for participants to first stool passage | 1 week
  The time needed for stool passage, in terms of hours

SECONDARY OUTCOMES:
Time for participants to resumption of feeding | 1 month
  time needed to resume feeding in terms of days
Time for participants to discharge from hospital after operation | 1 month
  in term of days
Presence of any complications in participants | 1 month
  any complication happened because of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University of Hong Kong, Hong Kong, Hong Kong